CLINICAL TRIAL: NCT02297165
Title: Efficacy Study of an Olfactory Stimulation Program in Relaxing Environment for the Recuperation of Autobiographical Memories in Anorexic Patients
Brief Title: Efficacy Study of an Olfactory Stimulation Program for the Recuperation of Autobiographical Memories in Anorexia
Acronym: OLFANOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P0028
Record Dates: First submitted 2014-11-04; First posted 2014-11-21 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2017-03

CONDITIONS: Anorexic
Keywords: anorexic; olfactory stimulation; autobiographical memories recovery
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program (Experimental): olfactory stimulation program
  Interventions: Behavioral: olfactory stimulation program
- Control (No Intervention): normal follow-up

INTERVENTIONS:
Behavioral: olfactory stimulation program — 8 individual sessions of olfactory stimulation at the rate of 2 sessions per week. 3 semi-directed interviews will be help (one at the beginning of the trial, the second 5 weeks later and the third at 6 month).
  For each session, patients have to smell two different odors (previously selected from a panel presented to the patient during first visits) and then they are invited to evoke memories and feelings related to each odor.
  Arms: Program

SUMMARY:
The purpose of this study is to estimate the impact of an olfactive stimulation, in relaxing environment, on the access at the autobiographical memories in anorexic patients.

ELIGIBILITY:
Inclusion Criteria:

* Eating disorders, anorexia (restrictive form or mixed) according to DSM IV-TR ( Diagnostic and Statistical Manual of Mental Disorders IV - Text Revision) criteria
* Patient hospitalized in a department of one of the inquiring centers for a minimal duration of 5 weeks
* French language ability
* Coverage by the social insurance
* Fully informed patient who consent to participate in the study

Exclusion Criteria:

* Major mental associated disorders (psychotic disorders, bipolar disorder, major depression), neurological disorders or addiction to substances
* Psychotropic treatment (with the exception of antidepressants, anxiolytics and sleeping drugs, if the treatment was started more than 30 days ago)
* Any disorder susceptible to alter the reasoning capacities, discernment or judgment
* Physically or psychologically unable to answer questionnaires

Ages: 13 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2017-09 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Proportion of reminded specific autobiographical memories (Autobiographical Memory Test (AMT) | After 5 weeks
  Autobiographical Memory Test (AMT) at inclusion and 5 weeks after

SECONDARY OUTCOMES:
Body mass index | first day of enrollment and 5 weeks after
  Evaluation of size and weight
Evaluation of the specific memories recovery stimulation on the emotional differentiation ability (Level of Emotional Awareness Scale (LEAS) | first day of enrollment and 5 weeks after
  Level of Emotional Awareness Scale (LEAS)
Evaluation of mental rumination (Cambridge Exeter Rumination Thinking Scale) | first day of enrollment and 5 weeks after
  Cambridge Exeter Rumination Thinking Scale
Evaluation of anxiety and depression (Hospital Anxiety and Depression Scale) | first day of enrollment and 5 weeks after
  Hospital Anxiety and Depression Scale
Evaluation of eating behaviors (Eating Disorder Inventory) | first day of enrollment and 5 weeks after
  Eating Disorder Inventory
Evaluation of history of abuse (Childhood Trauma Questionnaire) | first day of enrollment and 5 weeks after
  Childhood Trauma Questionnaire
Evaluation of cognitive avoidance strategies (Questionnaire of cognitive avoidance) | first day of enrollment and 5 weeks after
  Questionnaire of cognitive avoidance

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Dodin, Study Director — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No